CLINICAL TRIAL: NCT02979223
Title: Comparison the Efficacy Depending on the Order of the Sequential Combination Method Using Sodium Picosulfate and Magnesium Citrate (PMC) and PEG With Ascorbic Acid for Bowel Preparation (The Phase II Prospective Randomized Clinical Trial)
Brief Title: Combination Method Using Sodium Picosulfate and Magnesium Citrate and PEG With Ascorbic Acid for Bowel Preparation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Byung Chang KIM, Principle investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NCC2016-0166
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Bowel Preparation; Sodium Picosulfate and Magnesium Citrate; Polyethylene Glycol With Ascorbic Acid
MeSH Terms: interventions — picosulfate sodium; magnesium citrate; Polyethylene Glycols; Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PMC/PEG-Asc (Experimental): Picolyte 1 bottle/170cc at one day before colonoscopy, 7 PM. And then, Intake Coolprep 1L at the day of colonoscopy, 5 AM
  Interventions: Drug: sodium picosulfate and magnesium citrate, polyethylene glycol with ascorbic acid
- PEG-Asc/PMC (Active Comparator): Intake Coolprep 1L at one day before colonoscopy, 7 PM. And then, Intake Picolyte 1 bottle/170cc at the day of colonoscopy, 5AM
  Interventions: Drug: sodium picosulfate and magnesium citrate, polyethylene glycol with ascorbic acid

INTERVENTIONS:
Drug: sodium picosulfate and magnesium citrate, polyethylene glycol with ascorbic acid — sodium picosulfate and magnesium citrate and 2L polyethylene glycol with ascorbic acid are used as combination method.
  There is a difference in the order of intake between two group
  Other Names: Picosolution; Coolprep

SUMMARY:
The aim of this study is to compare the efficacy depending on the order of the sequential combination method using sodium picosulfate and magnesium citrate (PMC) and PEG with ascorbic acid for bowel preparation.

The investigators designed this study as a phase II prospective randomized parallel arm clinical trial. 71 participant will be enrolled in each group (142 in total).

The primary outcome is the efficacy of bowel preparation. secondary outcomes are tolerability, side effect of the drugs, polyp detection rate and adenoma detection rate.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-75 Patients who visited the outpatient clinic for colonoscopy Patients who agreed to participate in this study

Exclusion Criteria:

* pregnancy, breast feeding stage 3-5 chronic kidney disease (glomerular filtration rate < 60 mL/min/1.73m2), inability to maintain adequate fluid intake, pre-existing electrolyte disturbances, symptomatic congestive heart failure, recent (within < 6 months) symptomatic ischemic heart disease (unstable angina or myocardial infarction).

toxic megacolon active colitis Allergic to drug altered mental status Nausea and vomiting Hyperphosphatemia glucose-6-phosphate dehydrogenase deficiency Hereditary Phenylketonuria Patients with a history of colon surgery Abdominal operation within 6 months

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Successful bowel preparation (Excellent and Good in Aronchick bowel preparation score) | during colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Bun Kim, Dr, Principal Investigator — National Cancer Center, Korea
Locations (1):
- Bun Kim, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No